CLINICAL TRIAL: NCT06854432
Title: Multi-omics Approaches and Biometrological Analyses to Better Understand Androgenetic Alopecia: Exploratory Study
Brief Title: Assessment of Biological and Biometrological Parameters in Adult Subjects with Androgenetic Alopecia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: INTERALOPECIE
Record Dates: First submitted 2025-02-21; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Alopecia, Androgenetic; Healthy
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control subject group (Other)
  Interventions: Other: Biometrological measurements; Other: Biological sampling
- Subject group with androgenetic alopecia (Other)
  Interventions: Other: Biometrological measurements; Other: Biological sampling

INTERVENTIONS:
Other: Biometrological measurements — Measurements will be taken from the scalp: on the vertex and occiput areas.
Other: Biological sampling — Samples will be taken from the scalp: on the vertex and occiput areas.

SUMMARY:
Androgenetic alopecia is a chronic pathology affecting approximately 50% of men at 50 years old and is characterized by a progressive miniaturization of the hair follicle leading to a localized baldness.

Although it has been shown that testosterone metabolism plays a central role in this pathology, targeting this biological pathway is not fully efficient to treat androgenetic alopecia, suggesting that other factors are involved, notably factors linked to the perifollicular environment. Moreover, the very specific pattern of androgenetic alopecia is not yet fully understood: the occipital and lower temporal areas of the scalp are always preserved. Once the hair follicle has disappeared, it is not possible to make it grow back, it is then important to provide a treatment that slows down the progression of androgenetic alopecia at the earliest stage of the pathology, and that specifically targets the affected area.

The aim of this study is to better understand androgenetic alopecia pathophysiology by a multi-omic approaches and biometrological analysis, in the same study, on the local ecosystem of bald scalp areas and non-bald scalp areas of adult with androgenetic alopecia, compared to scalp of adult without androgenetic alopecia.

ELIGIBILITY:
Selection criteria:

Criteria related to the population:

* Male
* Subject aged between 30 and 50 years included

Criteria related to the scalp condition:

* Subject with hair length over 3 cm
* Subject presenting a negative pull test result

Specific for non-AGA group:

• Non-alopecic men with full head of hair with uniform scalp coverage (homogeneous hair density on the vertex, occiput, left and right parietal areas)

Specific for AGA group:

• Androgenetic alopecic men with progressive AGA for more than 5 years: stage between III to IV included according to the Hamilton's classification modified by Norwood

Non-selection criteria:

Criteria related to the population:

* Subject having received on study areas artificial UV exposure, excessive or prolonged exposure to natural sunlight within 2 months before the selection visit
* Subjects with frizzy hair

Criteria related to diseases:

* Subject having neoplastic disease (history of disease or disease on-going)
* Subject having severe acute progressive disease (infectious syndromes, inflammatory, COVID-19, acute fever...) occurred within the last 3 months before the selection visit liable to interfere with the study assessments
* Subject with iron deficiency on-going, not treated or treated for less than 3 months before the selection visit
* Subject having a dermatological condition, an acute, chronic or progressive disease or history of disease liable to interfere with the study data or considered by the investigator hazardous for the subject or incompatible with the study requirements

Specific for non-AGA group:

* Subject with any type of alopecia
* Subject with family history of androgenetic alopecia in the father with stage ≥ III according to the Hamilton's classification modified by Norwood

Specific for AGA group:

• Subject with non-androgenetic alopecia (Cicatricial alopecia, Alopecia aerata...)

Criteria related to procedures, treatments, products and/or hair care routine:

* Radiotherapy, chemotherapy
* Scalp surgery
* Systematic or local androgenetic alopecia treatment or product, taken or applied for more than 4 consecutive weeks during the last 6 months before the selection visit
* Any following hair care within the last 3 months before the selection visit: dyeing, bleaching, perm
* Systemic or local non-steroidal anti-inflammatory drug taken or applied on the scalp for more than 1 week during the last month (systematic NSAIDs) or 2 weeks (local NSAIDs) before the selection visit

Non-inclusion criteria:

Criteria related to the population:

* Subject having received on study areas artificial UV exposure, excessive or prolonged exposure to natural sunlight between selection and inclusion visit

Criteria related to the disease:

• Subject with any adverse event occurring between selection and inclusion visit liable to interfere with the study assessments

Criteria related to treatments and/or products:

• Any procedures, treatments, products and/or hair care taken, applied or performed between selection and inclusion visit liable to interfere with the study assessments

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Cutaneous pH measurement | baseline (Visit 1- Day 1)
Sebum quantification : by Lipidic Index (LI) - Sebumeter® | baseline (Visit 1- Day 1)
Skin elasticity : by determination of the mechanical property of the skin with a biomechanical device | baseline (Visit 1- Day 1)
Cutaneous hydratation : by Hydratation Index (IH) - DermaLab® | baseline (Visit 1- Day 1)
Cutaneous barrier integrity : by Trans-Epidermal Water Loss (TEWL) - Vapometer® | baseline (Visit 1- Day 1)
Lipidomic profile by mass spectroscopy (in-vivo measurements) | baseline (Visit 1- Day 1)
Lipidomic profile by sampling method (absorbent paper) | baseline (Visit 1- Day 1)
Microbiota analysis by sampling method (hair follicles) | baseline (Visit 1- Day 1)
Microbiota analysis by sampling method (swabs) | baseline (Visit 1- Day 1)
Metabolite analysis by sampling method (hair follicles) | baseline (Visit 1- Day 1)
Transcriptomic analysis by sampling method (hair follicles) | baseline (Visit 1- Day 1)
Transcriptomic analysis by sampling method (swabs) | baseline (Visit 1- Day 1)
Lipidomic profiles by sampling method (swabs) | baseline (Visit 1- Day 1)

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Research Center, Toulouse, France